CLINICAL TRIAL: NCT00003867
Title: Phase I Clinical Study of Every Three Week Irinotecan With Oral Capecitabine Given Twice Daily for Two Weeks Out of Three in Patients With Gastrointestinal and Other Solid Malignancies
Brief Title: Irinotecan and Capecitabine in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067031; P30CA013330 (NIH); AECM-1199903068; NCI-V99-1541
Record Dates: First submitted 1999-11-01; First posted 2004-02-16 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage IIIB breast cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage IV anal cancer; recurrent anal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; stage IIIA anal cancer; stage IIIB anal cancer; recurrent esophageal cancer; regional gastrointestinal carcinoid tumor; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; small intestine adenocarcinoma; small intestine lymphoma; small intestine leiomyosarcoma; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; unspecified adult solid tumor, protocol specific; newly diagnosed carcinoma of unknown primary; carcinoma of the appendix; recurrent carcinoma of unknown primary; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Breast Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Anus Neoplasms; Esophageal Neoplasms; Carcinoma, Hepatocellular; Gallbladder Neoplasms; Bile Duct Neoplasms; Appendiceal Neoplasms; Neoplasms, Unknown Primary | interventions — Capecitabine; Irinotecan

INTERVENTIONS:
Drug: capecitabine
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of irinotecan and capecitabine in treating patients who have solid tumors that have not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and toxic effects of irinotecan and oral capecitabine in patients with gastrointestinal or other solid tumors. II. Characterize the relationship at the recommended phase II dose between thymidine synthase and thymidine phosphorylase expression and tumor response and/or toxic effects in these patients.

OUTLINE: This is a dose escalation study. Patients receive oral capecitabine twice daily every twelve hours for 14 days, and IV irinotecan over 30 minutes once every 3 weeks beginning on day 1. Treatment continues for at least 2 courses in the absence of disease progression or unacceptable toxicity. The dose of capecitabine and irinotecan is escalated in cohorts of 3-6 patients until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 25-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed solid tumors, including but not limited to breast, gastrointestinal, and unknown primary cancer that is refractory to standard therapy or for which no standard therapy exists No known bone marrow involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 OR WBC at least 3,500/mm3 AND Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL No known Gilbert's syndrome No other significant hepatic disease requiring medication Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No significant cardiac disease requiring medication Other: Not pregnant or nursing Fertile patients must use effective contraception No other significant medical condition

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 2 weeks since prior colony stimulating factor and other cytokines active on bone marrow Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since mitomycin or nitrosoureas) No prior or concurrent irinotecan and fluorouracil therapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy No concurrent radiotherapy Surgery: Recovered from prior major surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-03 (Actual); Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Mani, MD, Study Chair — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Comprehensive Cancer Center, The Bronx, New York, United States

REFERENCES:
- [Result] Goel S, Jhawer M, Rajdev L, Hopkins U, Fehn K, Baker C, Chun HG, Makower D, Landau L, Hoffman A, Wadler S, Mani S. Phase I clinical trial of irinotecan with oral capecitabine in patients with gastrointestinal and other solid malignancies. Am J Clin Oncol. 2002 Oct;25(5):528-34. doi: 10.1097/00000421-200210000-00022. PMID 12393999